CLINICAL TRIAL: NCT01678833
Title: Neural Mechanistic Explanations for Differential Drug Abuse Treatment Outcomes
Brief Title: Understanding Drug Abuse Treatment Outcomes
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912480; 12-DA-N480
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-03-07

CONDITIONS: Drug Abuse/Dependence
Keywords: Drug Abuse/Dependence
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

Although some treatments for substance abuse are considered effective for some people who are drug dependent, many others do not benefit as much over time. Researchers are working to find out what characteristics predict treatment response. They also want to determine how to design treatments that are more effective for a greater number of substance abusers. This pilot study involves providing drug addicts with cognitive behavioral therapy (CBT), a treatment considered to be one of the most effective in reducing substance-abuse, to identify ways in which the brain works that may predict and explain treatment effects. A comparison group will be included that receives only standard psychotherapy or talk therapy. This approach will enable researchers to determine what factors might be interfering with favorable treatment outcomes and how to refine or develop new treatments that work well for more people.

Objectives:

- To identify individual characteristics which predict and explain the effects of CBT in people with opiate dependence.

Eligibility:

* Males between 18 and 60 years of age who are dependent on opioids (such as heroin).
* Participants must be willing to take buprenorphine and receive substance abuse counseling.

Design:

* Participants will be screened with a physical exam and medical history.
* Researchers will ask questions about participants ability to cope in certain situations, along with questions about drug use and lifestyle issues. These questions will be asked twice, before and after completing treatment.
* Participants will be placed into one of two groups. One group will have CBT twice a week for 8 weeks. The other group will have standard counseling twice per week. Both groups will take buprenorphine as part of the drug abuse treatment.
* Participants will have other tests during this study. They will have imaging studies to look at brain function. These studies will test thinking and decision making.

DETAILED DESCRIPTION:
OBJECTIVE:

The primary objective of this pilot study is to collect data for a NIH RO1 grant submission that aims to elucidate cognitive, emotional regulatory and neurobiological mechanisms that both moderate and mediate effects of cognitive behavioral therapy (CBT) in individuals with opiate dependence. CBT has proven moderately effective in treating substance abuse; however, significant variability in treatment outcomes remains. CBT curricula teach adaptive decision making and cognitive reappraisal skills to down-regulate emotional responses to drug-related cues, thereby promoting avoidance of drug use situations. A certain level of cognitive and emotion regulatory functioning is, however, required for assimilating and executing these skills which is often deficient in substance abusers. Consequently, many addicts cannot effectively process and act on CBT curriculum, leading to poor treatment outcomes. Tailoring interventions requires systematic investigation of neurobiological indicators that interfere with or promote favorable treatment responsivity.

The small pilot study outlined below will provide the feasibility and supportive data for a larger effort.

Aim 1: Moderation. Identify baseline ECF and emotion regulatory functions and their neural substrates that predict treatment variability in the form of: (a) program responsivity (e.g., treatment engagement, motivation, social competences) and (b) posttreatment outcomes (e.g., substance use frequency, days of continuous abstinence). Functional magnetic resonance imaging (fMRI) will be used during performance of tasks that measure ECF (decision-making; inhibitory control) and cognitive reappraisal of emotional cues to investigate the neuromodulatory role of PFC regions (e.g., OFC, ACC) on emotion (e.g., amygdala) and reward (e.g., ventral striatum) structures and autonomic activity.

Aim 2: Mediation. Determine whether change in these neurocognitive functions in response to CBT mediate intervention effects. Evidence suggests that CBT alters PFC and limbic function; such changes are associated with clinical outcomes in depression and anxiety. Similarly, in drug abusers, we predict treatment response will be associated with changes in neural activation patterns, ECF, and emotional regulation, and that little to no change will occur in those with relatively poorer outcomes.

Study Population: Participants will be 18 primary opioid dependent individuals between the ages of 18 and 60. These individuals will either be enrolled in NIDA Protocol 09-DA-N020, (Dr. Kenzie Preston, PI) or patients at the University of Maryland Medical Center outpatient substance abuse clinics (i.e., Alcohol and Drug Abuse Program (ADAP) or Outpatient Addiction Treatment Service (OATS) and are receiving buprenorphine.

DESIGN:

Study participants visit their treatment facility daily for buprenorphine and receive standard counseling as part of Protocol 09-DA-N020 or their treatment protocol at ADAP or

OATS. They will be screened by MMG for eligibility into the present study then randomly assigned to a TAU control group or a CBT group. This study consists of 3 assessment time points (baseline, midway, post-treatment) and 16 bi-weekly counseling visits (CBT or standard TAU counseling). Baseline assessments will consist of functional magnetic resonance imaging (fMRI) during performance of decision making, inhibitory control and emotional regulatory tasks. Questionnaires will be used to evaluate historical and current drug use, background and psychological traits, and other relevant factors. Those in the TAU group visit their treatment facility routinely for buprenorphine and standard counseling but will not receive CBT. The CBT group participants will undergo 8 weeks of CBT in the

Archway Clinic twice a week provided by a CBT clinician from Mountain Manor Treatment

Center who will be supervised by Dr. Marc Fishman, treatment director at MMTC; this CBT counseling will be in place of the TAU counseling they would be receiving as part of the parent protocol. Midway through CBT/TAU counseling, participants in this pilot study will be evaluated outside the scanner with the same cognitive tasks used in the scanner and questionnaires from baseline. After treatment completion, they will receive a post-treatment fMRI scan where they will perform the same tasks and questionnaires. Also, we will preliminarily assess mediation by examining variability in level of responsivity within the treatment group to determine whether this outcome is related to functional baseline characteristics and change over time. Expectations are that baseline features will predict intervention response and that these same characteristics will change over time in response to intervention in those with favorable outcomes.

OUTCOME MEASURES:

The focus of our outcome evaluation will be use of opioid (e.g., frequency, days of continuous abstinence, etc.), coping strategies, and change in lifestyle measures (e.g., employment, relationships, behavioral problems, treatment engagement).

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be eligible for inclusion in the study if they meet the following criteria:

1. Right-handed individuals between the ages of 18 and 60;
2. Good physical condition;
3. Participating and receiving buprenorphine treatment in protocol 09-DA-N020, a study being conducted in the NIDA Intramural Archway Clinic (Dr. Kenzie Preston, PI) in Baltimore, MD OR at outpatient treatment facilities at UMMC (ADAP or OATS);
4. Heroin or other opioid dependent;
5. Suitable for MRI scanning;

EXCLUSION CRITERIA:

Participants will be excluded from this study if they:

1. History of neurological illnesses including but not limited to CVA, CNS tumor, head trauma, MS or other demyelinating diseases, epilepsy, movement disorders, or migraine in treatment.
2. Are HIV infected.
3. Have deep vein thrombosis (DVT): Assessment tool: self report during H&P of thrombosis, family history of thrombosis, or a medical condition that may lead to a hypercoagulable state Rationale: Lying still for an hour (plus the mock scanning session) may be a risk for the development of DVT in persons with certain medical conditions. As such, persons with will be excluded.
4. Have current suicidal ideation.
5. Are unable to undergo MRI scanning due to metallic devices in the body including dental braces, claustrophobia or body morphometry.
6. Are currently using respiratory, cardiovascular or anticonvulsant medications that may interfere with the BOLD MRI signal.
7. Cognitively impaired;
8. Continued noncompliance (after the 3rd time) with respect to testing positive for illicit drugs or reporting caffeine use in the past 12 hours or alcohol use in the past 24 hours when they visit for their scanning sessions will lead to discontinuing their participation in the #480 protocol.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2012-07-19; Study Completion 2016-03-07

PRIMARY OUTCOMES:
The focus of our outcome evaluation will be use of opioid (e.g., frequency, days of continuous abstinence, etc.), coping strategies, and change in lifestyle measures (e.g., employment, relationships, behavioral problems, treatment engagement).

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (2):
- United States (2):
  - National Institute on Drug Abuse, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland

REFERENCES:
- [Background] Apodaca TR, Miller WR. A meta-analysis of the effectiveness of bibliotherapy for alcohol problems. J Clin Psychol. 2003 Mar;59(3):289-304. doi: 10.1002/jclp.10130. PMID 12579546
- [Background] Aharonovich E, Hasin DS, Brooks AC, Liu X, Bisaga A, Nunes EV. Cognitive deficits predict low treatment retention in cocaine dependent patients. Drug Alcohol Depend. 2006 Feb 28;81(3):313-22. doi: 10.1016/j.drugalcdep.2005.08.003. Epub 2005 Sep 19. PMID 16171953
- [Background] Aharonovich E, Brooks AC, Nunes EV, Hasin DS. Cognitive deficits in marijuana users: Effects on motivational enhancement therapy plus cognitive behavioral therapy treatment outcome. Drug Alcohol Depend. 2008 Jun 1;95(3):279-83. doi: 10.1016/j.drugalcdep.2008.01.009. Epub 2008 Mar 7. PMID 18329188